CLINICAL TRIAL: NCT04178603
Title: The COpenhagen-BOston-Sydney Study, The COBOS-study
Brief Title: Copenhagen, Boston, Sydney
Acronym: COBOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Pfizer (Industry); University of Sydney (Other)
Responsible Party: Principal Investigator, Professor Jorgen FP Wojtaszewski, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: COBOS
Record Dates: First submitted 2019-11-18; First posted 2019-11-26 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-04

CONDITIONS: Insulin Resistance; Insulin Sensitivity; Type 2 Diabetes
Keywords: Exercise; Insulin Resistance; Type 2 Diabetes; Glucose Uptake; Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Lean control subjects and obese insulin resistant subjects undergo two different trials (trial A and B). Trial A aims to investigate the effect of acute exercise and 2 hours recovery. Trial B aims to investigate insulin sensitivity for glucose uptake in recovery from exercise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Exercise Trial (Experimental): Lean control subjects and insulin resistant subjects perform an acute bout of one-legged knee-extensor exercise. Glucose metabolism is investigated before exercise (basal), during exercise and for 120 min of recovery.
  Interventions: Other: Exercise, insulin infusion
- Insulin Sensitivity post Exercise (Experimental): Lean control subjects and insulin resistant subjects perform an acute bout of one-legged knee-extensor exercise and insulin action is investigated 4 hours after cessation of exercise. Insulin action is investigated by a 120 min euglycemic-hyperinsulinemic euglycemic clamp.
  Interventions: Other: Exercise, insulin infusion

INTERVENTIONS:
Other: Exercise, insulin infusion — Trial A: Acute one-legged exercise Trial B: Insulin infusion 4 hours after one-legged exercise

SUMMARY:
The study investigates the regulation of muscle glucose utilization during exercise and enhanced insulin sensitivity in recovery from exercise.

This will be investigated in lean control subjects and obese insulin resistant subjects.

DETAILED DESCRIPTION:
The subjects will perform two trials (trial A and B).

Trial A: During trial A the study subject will eat a morning meal at 6:00 a.m. corresponding to 5% of the daily energy requirements and will arrive at the research laboratory at 8:00 a.m. It is requested that the study subject will arrive in a car or with public transportation. After arrival the study subject will rest for 1 hour and at that time catheters are inserted in both femoral veins and the femoral artery in one of the legs. At 9:00 a.m. the study subjects will perform one-leg knee extension exercise for 1 hour at an intensity of 80% of maximal work capacity. In this work protocol there are inserted 3 intervals of 5 minutes duration where the study subject works at 100% of maximal intensity with the purpose of securing a full activation/recruiting of all muscle fibers. Muscle biopsies from the m. vastus lateralis muscle in both legs will be taken before (at 8.45 a.m.), immediately after (at 10:00 a.m.) and 2 hours after conclusion of exercise (at 12:00 p.m.) (in total of 6 biopsies). Pulmonary oxygen uptake is measured with the use of an online system before, during and after exercise and is used for determination of substrate metabolism. Blood samples from the femoral veins in both legs and the femoral artery in one of the legs are drawn before (at 8:20 a.m., 8:40 a.m. and 9:00 a.m.), during exercise (at 9:20 a.m., 9:40 a.m. and 10:00 a.m.) and during the recovery period after exercise (at 10:10 a.m., 10:30 a.m., 11:00 a.m., 11:30 a.m. and 12:00 p.m.). At the same time blood flow is measured in the femoral arteries in both legs with the use of Doppler technique. Determination of arteriovenous difference (AV difference) by simultaneous measurement of blood flow enables us to calculate skeletal muscle glucose uptake and uptake/release of relevant substances (proteins, peptides and metabolites etc.). The experimental part of trial A is completed at 12:00 p.m. The study subject will be given food and drink and will be observed for one hour before they may leave the research laboratory.

Trial B: During test trial B the study subjects will eat a morning meal at 6:00 a.m. corresponding to 5% of the daily energy requirements and will arrive at the research laboratory at 8:00 a.m. It is requested that the study subject will arrive in a car or with public transportation.

During trial B the study subjects will perform the same one-leg knee extension exercise protocol as in trial A. At 9:00 a.m. the study subject starts performing one-leg knee extension exercise for 1 hour at 80% of maximal work capacity with 3 intervals of 5 minutes duration where the load is at 100% of maximal work capacity. This work protocol ensures full activation/recruiting of all muscle fibers. After the kicking exercise is completed the study subject will rest in supine position for 6 hours. At the beginning of this resting period catheters are inserted in the femoral veins in both legs and in the femoral artery in one leg. Also catheters are inserted in each forearm vein (antecubital veins) for intravenous infusion of insulin, glucose and stable 13C(u)-glucose. Intravenous infusion of 13C(u)-glucose is started 2 hours after conclusion of exercise in order to achieve a 10% enrichment of blood glucose. 4 hours after cessation of exercise a hyperinsulinemic euglycemic clamp of 120 minutes duration is started. This implies intravenous infusion of insulin and glucose for 120 minutes in order to determine insulin sensitivity for glucose uptake and metabolism of glucose. The clamp is started with a bolus injection of insulin (9.0 mU/kg) followed by a constant infusion (1.42 mU/kg/min). Simultaneously glucose infusion rate will be adjusted so that euglycemia is maintained. Immediately before, after 30 minutes and after 120 minutes of insulin infusion a muscle biopsy is taken from the vastus lateralis muscle in both legs (a total of 6 biopsies). Blood samples from both femoral veins and one femoral artery are taken before (at 12:00 p.m., 12:30 p.m., 1:00 p.m., 1:30 p.m. and 2:00 p.m.) and during (at 2:15 p.m., 2:30 p.m., 2:45 p.m., 3:00 p.m., 3:15 p.m., 3:30 p.m., 3:45 p.m. and 4:00 p.m.) the hyperinsulinemic euglycemic clamp. Simultaneously blood flow is measured in both femoral arteries with use of Doppler technique. Determination of arteriovenous difference (AV difference) by simultaneous measurement of blood flow enables us to calculate glucose uptake and uptake/release of relevant substances (proteins, peptides and metabolites etc.). Indirect calorimetry for determination of whole body metabolism is measured concomitantly, starting 2 hours after conclusion of exercise. The experimental part of trial B is concluded at 4:00 p.m. The study subjects receive food and drink and are observed for one hour before they may leave the research laboratory.

Muscle biopsies and blood samples from trial A and B are stored in a locked -80ºC freezer. Muscle samples and blood samples will subsequently be used for miscellaneous analyses described under background.

The trials (A and B) will be carried out in a randomized order and will be separated by a minimum of 14 days.

ELIGIBILITY:
Inclusion Criteria for Study Subjects

* Healthy persons (no known disease) without diabetes in the family
* No use of medications
* Non-smokers
* Men
* Age 25-40 years
* Physical activity level (VO2peak) between 30-50 mL O2/min/kg

Specific for the persons of normal weight:

* BMI between 18.0 and 25.0
* HOMA-IR ≤ 1.5
* Glucose tolerant (intact response in relation to oral glucose tolerance test, OGTT)
* Without metabolic syndrome (defined by the International Diabetes Federation in 2006)

Specific for the persons with overweight and insulin resistance:

* BMI between 28.0 and 35.0
* HOMA-IR ≥ 2.2
* Glucose tolerant (intact response in relation to OGTT)

Exclusion criteria

* Women
* Elevated blood pressure (systolic above 140 mmHg, diastolic above 90 mmHg).
* Persons who show signs of metabolic diseases, hematologic diseases, reduced liver function or other signs of disease that may affect the outcome of the study or the study subject's wellbeing will be excluded.

Exclusion after Inclusion

* If disease appears or is identified and/or a need for medication arises after inclusion but before initiation of the study.
* Disease during conclusion of the study

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Muscle glucose uptake during exercise and enhanced insulin sensitivity in recovery from exercise. | Through study completion, an average of 1 year.
  Muscle glucose uptake during exercise and during insulin stimulation in recovery from exercise (insulin sensitivity) will be determined based on the the Fick principle. Thus, arterio-venous difference (av difference) in blood glucose will be multiplied by arterial leg blood flow.

SECONDARY OUTCOMES:
Posttranslational modification of proteins in muscle biopsies. | 5 years
  The obtained muscle samples will be subjected to mass spectrometry analysis. This measurement shows posttranslational modification that regulates protein function.

OTHER OUTCOMES:
Changes in content of metabolites in muscles and blood plasma as a result of exercise and during subsequent insulin stimulation. | 5 years
  Concentration of several hundreds of metabolites in glucose, lipid and protein metabolism will be analyzed by mass spectrometry and liquid chromotography.
Changes in gene-expression in muscle as a result of exercise and during subsequent insulin stimulation. | 5 years
  Gene-expression in muscle samples will be measured by RNA.sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Exercise, Nutrition and Sports, Faculty of Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No